CLINICAL TRIAL: NCT04070417
Title: Lifestyle Medicine for Depression: A Pilot Randomized Controlled Trial
Brief Title: Lifestyle Medicine for Depression 2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Melbourne (Other); University of Western Sydney (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY007
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Depression
Keywords: Depression; Lifestyle Medicine
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Lifestyle Medicine Group
  Interventions: Behavioral: Lifestyle Medicine
- CAU Group (No Intervention): Care-As-Usual Group

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Lifestyle intervention with components including physical activity, diet, relaxation/mindfulness, sleep and socialisation
  Arms: Treatment Group

SUMMARY:
This study will examine the feasibility and efficacy of lifestyle medicine for the enhancement of psychological wellness in adult. The main components of lifestyle intervention typically include physical activity, diet, relaxation/mindfulness, sleep and socialisation. These components are weaved with psychological elements such as stress management, cognitive restructuring, motivational interviewing, and goal setting strategies that are led by clinical psychologists. While lifestyle medicine has been recognised for centuries a a mean to improve physical health, the field of lifestyle medicine in the context of mental health is still in its infancy. Nevertheless, there is increasing evidence demonstrating the efficacy of individual components of lifestyle medicine (e.g. diet, physical activities, and sleep) on mood and stress management. With a well-researched lifestyle medicine programme adopted from Australia, the research team of the Chinese University of Hong Kong has customised the intervention protocol to fit the Chinese culture.

The investigators aim to examine the effectiveness of an integration of multiple lifestyle adjustments on depression from a holistic body-mind perspective.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged ≥ 18 years;
* Cantonese language fluency;
* Patient Health Questionnaire (PHQ-9) score ≥ 10; and
* Willingness to provide informed consent and comply with the trial protocol

Exclusion Criteria:

* Pregnancy;
* Have suicidal ideation with PHQ-9 item 9 score ≥ 2 (referral information to professional services will be provided to those who endorsed items on suicidal ideation);
* Using medication or psychotherapy for depression;
* Having unsafe conditions and are not recommended for physical activity or a change in diet by physicians; and
* Have major psychiatric, medical or neurocognitive disorders that make participation infeasible or interfere with the adherence to the lifestyle intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, 1-week post-treatment and 12-week post treatment
  The PHQ-9, a 9-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in the Depression Anxiety Stress Scales (DASS-21) | Baseline, 1-week post-treatment and 12-week post treatment
  DASS-21 is a 21-items scales, comprises of three sub-scales which measures the negative emotional states of depression, anxiety, and stress, over the past week. The DASS is based on a dimensional rather than a categorical conception of psychological disorder, thus it has no direct implications for the allocation of patients to discrete diagnostic categories. However, recommended cutoff scores for conventional severity labels (normal, moderate, severe) are given in the DASS Manual.
Change in the Insomnia Severity Index (ISI) | Baseline, 1-week post-treatment and 12-week post treatment
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, 1-week post-treatment and 12-week post treatment
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | Baseline, 1-week post-treatment and 12-week post treatment
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the Sheehan Disability Scale (SDS) | Baseline, 1-week post-treatment and 12-week post treatment
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline and 1-week post-treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong